CLINICAL TRIAL: NCT02375048
Title: Randomized Study on Postmenopausal Women With Early Stage Breast Cancer: Adjuvant Hypofractionated Whole Breast Irradiation (WBI) Versus Accelerated Partial Breast Irradiation (APBI)
Brief Title: Randomized Study on Postmenopausal Women With Early Stage Breast Cancer: WBI Versus APBI
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: number of enrollments not reached in the estimated time
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Principal Investigator, Michele Tedeschi, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1288
Record Dates: First submitted 2015-02-13; First posted 2015-03-02 (Estimated); Last update posted 2018-10-24 (Actual); Status verified 2018-10

CONDITIONS: Cancer of Breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Hypofractionated WBI (Active Comparator): Patients treated with hypofractionated Whole Breast Irradiation received Simultaneous Integrated Boost irradiation of the whole breast and surgical bed at two different dose levels using external intensity - modulated radiotherapy (VMAT RA).
  Interventions: Radiation: Hypofractionated WBI
- Accelerated Partial Breast Irradiation (Experimental): Patients treated with Accelerated Partial Breast Irradiation received the irradiation on surgical bed using external intensity - modulated radiotherapy (VMAT RA).
  Interventions: Radiation: Accelerated Partial Breast Irradiation

INTERVENTIONS:
Radiation: Hypofractionated WBI — Dose prescription was 40.5 Gy to PTVWB and 48.0 Gy to PTVboost in 15 fractions over 3 weeks, with simultaneous integrated boost delivering 2.7 and 3.2Gy/fraction for each PTV respectively. Daily image guided radiotherapy (IGRT) were generated before each treatment session in each patient to verify the set-up.
  Arms: Hypofractionated WBI
Radiation: Accelerated Partial Breast Irradiation — APBI was delivered at a dose of 30 Gy in five 6-Gy/day fractions over 10 days (every other day) with IGRT at each treatment.
  Arms: Accelerated Partial Breast Irradiation

SUMMARY:
Selected patients with early stage breast cancer undergone conservative surgery were randomized in two arms: Hypofractionated Whole Breast Irradiation versus Accelerated Partial Breast Irradiation.

DETAILED DESCRIPTION:
Patients treated with Hypofractionated Whole Breast Irradiation (WBI) received SIB irradiation of the whole breast and surgical bed at two different dose levels. Dose prescription was 40.5 Gy to PTVWB and 48.0 Gy to PTVboost in 15 fractions over 3 weeks, with simultaneous integrated boost delivering 2.7 and 3.2Gy/fraction for each PTV respectively. Daily image guided radiotherapy (IGRT) were generated before each treatment session in each patient to verify the set-up.

Accelerated Partial Breast Irradiation (APBI) using external intensity -modulated radiotherapy (VMAT RA) was delivered at a dose of 30 Gy in five 6-Gy/day fractions over 10 days (every other day) with IGRT at each treatment.

ELIGIBILITY:
Inclusion Criteria:

* 55< Age <70
* Tumor size ≤ 2 cm
* pN0 (SN biopsy or ALND)
* ER/PgR positive
* Margins > 5 mm (either at initial surgery or at re-excision)
* Clips placed in the surgical bed (minimum of 4 clips)
* Unicentric only
* No lymphovascular invasion
* Any grade
* No extensive intraductal component (>25%)
* Written informed consent

Exclusion Criteria:

* Prior thoracic radiation therapy
* Oncoplastic surgery / No clips in the surgical bed
* Multicentric cancer
* Autoimmune disease, vasculitis, collagenopathy or scleroderma that may predispose to late sequelae

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2015-01-19 (Actual); Primary Completion 2018-02-01 (Actual); Study Completion 2018-02-01 (Actual)

PRIMARY OUTCOMES:
Toxicity will be measured with CTCAE v.4.0 | ten years
Cosmesis will be measured with Harvard scale | ten years

SECONDARY OUTCOMES:
Rate of Local Control | ten years
Disease Free Survival | ten years
Overall Survival | ten years
Quality of Life Questionnaire | ten years

CONTACTS AND LOCATIONS:
Overall Officials: Marta Scorsetti, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milano, Italy